CLINICAL TRIAL: NCT03779165
Title: R Wave Sensing After Radiofrequency Ablation of Ventricular Tachycardia Substrate in Patients With Structural Heart Disease
Brief Title: R Wave Sensing After VT Ablation
Acronym: RASA-VT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital Sestre Milosrdnice (Other)
Responsible Party: Principal Investigator, Ivan Zeljkovic, Principal Investigator, University Hospital Sestre Milosrdnice
Other Study IDs: ZAPSA01; UTN U1111-1223-2331 (Other: Universal Trial Number - World Health Organization)
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Tachycardia, Ventricular; Catheter Ablation; Follow-Up Studies; Electrodes
Keywords: ventricular tachycardia; R wave; sensing; radiofrequency ablation; follow-up
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sustained, monomorphic ventricular tachycardia (VT) is most commonly encountered in patients with structural heart disease, usually with ischemic aetiology. It has been proven that repeated episodes of sustained VT contribute to the mortality of patients with structural heart disease. These patients are usually implanted with implantable cardioverter defibrillator without (ICD) or with cardiac resynchronisation therapy (CRT-D). According to the current guidelines 3D mapping with radiofrequency (RF) ablation of the tachycardia substrate is an established therapeutic option. As part of the clinical follow-up of patients implanted with cardiac implantable electronic devices (CIED), CIED function parameters are monitored every 6 months, which is always done before and after any procedure involving RF ablation. Furthermore, a transient drop of R wave sensing has been demonstrated after the atrioventricular (AV) node ablation in patients with single-chamber pacemakers and fast atrial fibrillation. The aim of this study is to assess the change in R wave sensing after the RF ablation of VT substrate.

This study will be performed as a clinical, prospective, multi-centre, observational cohort study with a structured follow-up period of 12 months. All consecutive patients with sustained VT implanted with ICD or CRT-D undergoing RF ablation procedure of myocardial substrate, who are able to understand and sign informed consent, will be enrolled. Primary objective is a R wave sensing drop > 30% after VT substrate ablation procedure. Recruiting should not exceed 12 months with the minimal follow-up period of 12 months (24 months in total). Standardized statistical methods and test will be done using SPSS Software Version 22.0 or newer.

This unique study offers the possibility to show the impact of RF ablation on short-term and long-term R wave sensing change assessed by ICD or CRT-D's ventricle electrode in patients with sustained VT and structural heart disease undergoing ablation procedure. This observational data is needed to further refine the treatment of these patients and to prevent possible ICD/CRT-D dysfunction which could endanger this patient population.

DETAILED DESCRIPTION:
Sustained, monomorphic ventricular tachycardia (VT) is most commonly encountered in patients with structural heart disease, usually with ischemic aetiology. It has been proven that repeated episodes of sustained VT contribute to the mortality of patients with structural heart disease. These patients are usually implanted with implantable cardioverter defibrillator without (ICD) or with cardiac resynchronisation therapy (CRT-D) as part of sudden cardiac death (SCD) prevention and have had activation of the device due to the sustained VT episodes. According to the current guidelines 3D mapping with radiofrequency (RF) ablation of the tachycardia substrate is an established therapeutic option. As part of the clinical follow-up of patients implanted with cardiac implantable electronic devices (CIED), including ICDs and CRT-Ds, function parameters are monitored every 6 months. The same check-up is done before and after any procedure involving RF ablation. Furthermore, a transient drop of R wave sensing has been demonstrated after the RF ablation of the atrioventricular (AV) node in patients with uncontrollable fast atrial fibrillation implanted with single-chamber pacemakers. The above mentioned have not been studied yet in patients ablated due to sustained VT. Hence, the aim of this study is to assess the change in R wave sensing after the RF ablation of VT substrate in patients with structural heart disease.

This study will be performed as a clinical, prospective, multi-centre, observational (analytic, longitudinal) cohort study with patient enrolment in 4 electrophysiology centres in Croatia and Switzerland and a structured follow-up period of 12 months.

All consecutive patients with sustained VT implanted with ICD or CRT-D undergoing RF ablation procedure of myocardial substrate, who are able to understand and sign informed consent, will be enrolled.

Exclusion criteria:

* Patients with combined mechanical aortic and mitral valve prostheses
* Patients with RF ablation of VT done in the last 12 months
* Patients with known damaged ICD/CRT-D electrode or battery
* Patients undergoing VT ablation who have not been implanted with ICD or CRT-D
* Patients not willing or able to undergo clinical follow-up of ICD/CRT-D device
* Patients with life expectancy < 1 year
* Not able to understand or willing to sign informed consent
* Age < 18 years Primary objective is a R wave sensing drop > 30% after VT substrate ablation procedure.

Specific (secondary) end-points:

* incidence of VT recurrence after the ablation procedure;
* risk factors for R wave sensing drop (> 30%) after the RF ablation of VT substrate;
* time needed for R wave sensing recovery after the RF ablation procedure. Recruiting should not exceed 12 months with the minimal follow-up period of 12 months (24 months in total).

The risk categorisation of the study was done and the study was awarded a risk category A.

Sample size was chosen according to annual procedure volumes in Croatia and Switzerland. In addition, it is confirmed by power test (number needed to recruit: 52). Recruiting should not exceed 12 months. Categorical variables will be presented by contingency tables in absolute values and percentages. Categorical variables will be compared by the chi-square with Yates corrections or Fisher's exact test. Continuous data will be expressed as means and standard deviations or median with corresponding interquartile range. The differences in quantitative variables will be tested by Mann-Whitney U-test (non-parametric test for independent samples). Logistic regression will be used to analyse the association between all variables of interest and the R wave sensing drop. Multivariate logistic regression will be used to adjust for confounding factors. Predictors of the R wave sensing drop will be assessed in a univariate and multivariate Cox proportional hazards model. The statistical analysis will be done using SPSS Software Version 22.0 or newer (IBM SPSS Statistics, New York, USA).

This unique study offers the possibility to show the impact of RF ablation on short-term and long-term R wave sensing change assessed by ICD or CRT-D's ventricle electrode in patients with sustained VT and structural heart disease undergoing ablation procedure. This observational data is needed to further refine the treatment of these patients and to prevent possible ICD/CRT-D dysfunction which could endanger this patient population. Despite a high number of cohort registries for cardiovascular diseases (e.g. Danish heart registry, ORBIT-AF, GARFIELD AF registry, Swiss AF registry), there are scarce data on patients with structural VT and no data regarding R wave sensing changes influenced by RF energy application in ventricles. In addition, this could influence obligatory rhythm-monitoring duration and consequently hospitalization duration of patients with VT undergoing RF ablation procedures. Apart from the above mentioned, in those patients with non-optimal preprocedural R wave sensing, this could mean contraindication for procedure or having the need to do postprocedural defibrillation testing. It is likely, that data from our study will lead to future changes in periprocedural planning and modalities.

This study will be conducted in compliance with the current version of the Declaration of Helsinki, the ICH-GCP or ISO EN 14155 (as far as applicable) as well as all national legal and regulatory requirements. According to ethical regulations, the study plan with the proposed participant information and consent form as well as other project-specific documents will be submitted to Ethic committee of the participating centres.

ELIGIBILITY:
Inclusion Criteria:

* patients with recurrent, sustained ventricular tachycardia
* patients implanted with implantable cardioverter defibrillator (ICD) or cardiac resynchronization therapy cardioverter defibrillator (CRT-D)
* patients planned for 3D mapping and radiofrequency ablation of ventricular tachycardia myocardial substrate
* patients who are able to understand and sign informed consent

Exclusion Criteria:

* Patients with combined mechanical aortic and mitral valve prostheses
* Patients with RF ablation of VT done in the last 12 months
* Patients with known damaged ICD/CRT-D electrode or battery
* Patients undergoing VT ablation who have not been implanted with ICD or CRT-D
* Patients not willing or able to undergo clinical follow-up of ICD/CRT-D device
* Patients with life expectancy < 1 year
* Not able to understand or willing to sign informed consent
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with structural heart disease (ischemic and non-ischemic aetiology) implanted with implantable cardioverter defibrillator (ICD) or cardiac resynchronization therapy cardioverter defibrillator (CRT-D) and recurrent, sustained, monomorphic ventricular tachycardia, who are, according to their cardiologist, planned for 3D mapping and radiofrequency ablation of ventricular tachycardia myocardial substrate.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
R wave sensing change | immediately after the ablation procedure
  R wave sensing drop > 30% after RF ablation of VT substrate in left and/or right ventricle assessed by ventricular electrode of the CIED

SECONDARY OUTCOMES:
R wave sensing change 24h follow-up | 24 hours after ablation procedure
  R wave sensing drop > 30% after RF ablation of VT substrate in left and/or right ventricle assessed by ventricular electrode of the CIED
R wave sensing change 3-6 month follow-up | 3-6 months after ablation procedure
  R wave sensing drop > 30% after RF ablation of VT substrate in left and/or right ventricle assessed by ventricular electrode of the CIED
R wave sensing change 9-12 month follow-up | 9-12 months after the ablation procedure
  R wave sensing drop > 30% after RF ablation of VT substrate in left and/or right ventricle assessed by ventricular electrode of the CIED
Incidence of VT recurrence after the ablation procedure | 12 months after the ablation procedure
  Assessing the VT recurrence after the ablation procedure by ICD or CRT-D interrogation adn function testing
Risk factors for R wave sensing change after the RF ablation of VT substrate | 12 months
  assessing risk factors for R wave sensing drop after the RF ablation of VT substrate

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Zeljkovic, MD, Principal Investigator — University Hospital Sestre Milosrdnice
Locations (4):
- Croatia (2):
  - University Hospital Rijeka, Rijeka
  - University Hospital Sestre milosrdnice, Zagreb
- Switzerland (2):
  - University Hospital Basel, Basel
  - University Hospital Bern, Bern

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Darrat YH, Agarwal A, Morales GX, Thompson J, Abdel-Latif A, Waespe K, DI Biase L, Natale A, Patwardan A, Elayi CS. Radiofrequency and Cryo-Ablation Effect on Transvenous Pacing and Defibrillatory Lead Integrity: An In Vitro Study. J Cardiovasc Electrophysiol. 2016 Aug;27(8):976-80. doi: 10.1111/jce.13007. Epub 2016 Jun 14. PMID 27138905
- [Result] Priori SG, Blomstrom-Lundqvist C, Mazzanti A, Blom N, Borggrefe M, Camm J, Elliott PM, Fitzsimons D, Hatala R, Hindricks G, Kirchhof P, Kjeldsen K, Kuck KH, Hernandez-Madrid A, Nikolaou N, Norekval TM, Spaulding C, Van Veldhuisen DJ; Task Force for the Management of Patients with Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death of the European Society of Cardiology (ESC). 2015 ESC Guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death: The Task Force for the Management of Patients with Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death of the European Society of Cardiology (ESC)Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC). Europace. 2015 Nov;17(11):1601-87. doi: 10.1093/europace/euv319. Epub 2015 Aug 29. No abstract available. PMID 26318695